CLINICAL TRIAL: NCT00776724
Title: A Randomized Phase III Study of Docetaxel/ Epirubicin Versus Tailored Regimens as Neoadjuvant Chemotherapy for Stage II/III Breast Cancer With Tumor Size More Than 2 cm
Brief Title: Tailored Neoadjuvant Chemotherapy for Stage II/III Breast Cancer With Tumor Size More Than 2 cm
Acronym: TaiNAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200803006M
Record Dates: First submitted 2008-10-19; First posted 2008-10-21 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Chemotherapy
Keywords: breast ca; phase III; Tailored neoadjuvant chemotherapy; stage II/III
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): docetaxel-epirubicin for 4 cycles before surgery
  Interventions: Drug: Taxotere , Epirubicin
- 2 (Experimental): Tailored regimens, base on immunohistochemical study of the tumor biopsy tissue, for 4 cycles before surgery.
  Interventions: Drug: E-HDFL,EP,TE,N-HDFL,NP,T-HDFL,TP

INTERVENTIONS:
Drug: Taxotere , Epirubicin — Taxotere 70 mg/m2 1hr iv infusion / Epirubicin 90 mg/m2 (TE) iv infusion on day 1.
  Arms: 1
Drug: E-HDFL,EP,TE,N-HDFL,NP,T-HDFL,TP — Tau+ topo II+ ERCC1+ : Epi 45mg/m2 iv / 5FU 2000mg/m2 + Lv 300mg/m2 24 hrs infusion, day 1 and 8.
  Tau+ topo II+ ERCC1- : Epi 45mg/m2 iv/ Cis 35mg/m2 24 hrs iv infusion day 1 and 8.
  Tau+ topo II- ERCC1+ : Vin 25mg/m2 iv / 5FU 2000mg/m2 + Lv 300mg/m2 24 hrs infusion, day 1 and 8.
  Tau+ topo II- ERCC1- : Cis 35mg/m2 24 hrs infusion / Vin 25mg/m2 iv day 1 and 8.
  Tau- topo II+ ERCC1+ : Docetaxel 70 mg/m2 / Epirubicin 90 mg/m2 on day 1.
  Tau- topo II+ ERCC1- : Docetaxel 70 mg/m2 / Epirubicin 90 mg/m2 on day 1.
  Tau- topo II- ERCC1+ : Tax 35mg/m2 1hr infusion / 5FU 2000mg/m2 + Lv 300mg/m2 24 hrs infusion, day 1 and 8.
  Tau- topo II- ERCC1- : Tax 35mg/m2 1hr infusion / Cis 35mg/m2 24 hrs infusion day 1 and 8.
  Arms: 2

SUMMARY:
This is a multi-center randomized phase III trial. The purpose is to evaluate and compare the pathological complete response (pCR) rates after neoadjuvant chemotherapy with tailored chemotherapeutic regimens or standard chemotherapy for stage II/III breast cancer with tumor size more than 2 cm.

DETAILED DESCRIPTION:
This is a multicenter randomized phase III trial. The purpose is to evaluate and compare the pathological complete response (pCR) rates after neoadjuvant chemotherapy with tailored chemotherapeutic regimens or standard chemotherapy for stage II/III breast cancer with tumor size more than 2 cm.

For primary operable breast cancer, neoadjuvant chemotherapy is one of standard options. Pathological complete response (pCR) was associated with significantly improved long-term disease free and overall survival. Anthracycline/taxane-based chemotherapy regimens have been studied extensively in prospective trials and are the most frequently prescribed treatments in patients with breast cancer as neoadjuvant chemotherapy. Regimens that have been tested in large multicenter phase III trials and yielded pCR rates of at around 15% and up to 20% after 6 cycles of chemotherapy. Recent evidences have showed that the expression of several proteins in the tumor samples such as tau, topoisomerase II alpha (topo II), and ERCC1 can predict the tumor response to taxanes, anthracyclines, and platinums, respectively. We hypothesized that select chemotherapeutic agent according the expressions of drug sensitivity predictive biomarkers from patient's tumor sample may improve the efficacy of breast cancer treatment.

In this randomized phase III trial, TE (Docetaxel/ epirubicin) will be given in control arm since it is a highly active regimen for breast cancer. In the Tailored chemotherapy arm, 7 different combination chemotherapy regimens that containing 2 drugs among taxotere, epirubicin, cisplatin, vinorelbine, and 5FU, will be given according to the expressions of tumor biomarkers. The doses and schedules of those regimens are selected according published 1st line protocols for breast cancer. The primary endpoint is the pCR rate. After 4 cycles of neoadjuvant chemotherapy, under the assumption of pCR rate of 15% in TE arm, to achieve 80% power at the 5% level (one side) of significance for the detection of a 15% increase of pCR rate in tailored regimen arm, 134 patients in either arm should be included in the study. If a 10% drop-out rate and multi-center study variation effect are considered, totally 316 patients will be required.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive, but non-inflammatory, breast carcinoma, with stage II or III disease (AJCC 7th ed)
* And, tumor size more than 2 cm in greatest diameter measured by estimated by CT scan or MRI
* Documented Her2/neu negative , including score 0, 1+, or 2+ by immunohistochemistry
* No prior radiotherapy, hormonal therapy or chemotherapy for invasive breast cancer
* Performance status of ECOG 0, 1,
* Female with age older than 20 years
* Laboratory parameter

  * Absolute neutrophil count (ANC) ≧1500/mm3
  * Total bilirubin ≦2.0 times the upper limit of normal (ULM)
  * AST or ALT ≦2.5 times the upper limit of normal (ULM)
  * Platelets ≧100,000/mm3
  * Serum creatinine ≦1.5 x ULM
  * Fasting triglyceride ≧ 70 mg/dL
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Evidence of metastatic breast cancer or inflammatory breast cancer
* Bilateral breast cancer, metaplastic carcinoma, or mucinous carcinoma
* Known allergy to any of the study drugs or to agents containing Cremophor.
* Serious intercurrent infections or medical illnesses that are uncontrolled or the control of which may be jeopardized by this therapy
* Psychiatric disorders or other conditions regarding the subject incapable of complying with the requirements of the protocol
* Evidence of baseline sensory or motor neuropathy
* Pregnant or breast feeding women
* Previous or current systemic malignancy with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ with a disease-free interval of at least 5 years

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-05-29 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the pathological complete response (pCR) rates | operation after 4 cycles of neoadjuvant chemotherapy with tailored chemotherapeutic regimens or TE

SECONDARY OUTCOMES:
To evaluate the overall clinical response rate | after 4 cycles of neoadjuvant chemotherapy with tailored chemotherapeutic regimens or TE

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, M.D., Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital; Chiun-Sheng Hunag, MD,PhD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan